CLINICAL TRIAL: NCT05034822
Title: A Maximum Use (MUsT) Pediatric Study of 1.5% Ruxolitinib Cream in Children (Ages ≥ 2 Years to < 12 Years) With Atopic Dermatitis
Brief Title: Study of Ruxolitinib Cream in Children With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: Innovaderm Research (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 18424-109
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Atopic Dermatitis
Keywords: pediatric; Atopic dermatitis; ruxolitinib cream; maximum use; open label
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Masking Description: Images will be taken and masked for privacy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib cream (Experimental): ruxolitinib 1.5% cream will be applied twice daily to all areas of the skin affected by AD
  Interventions: Drug: Ruxolitinib cream

INTERVENTIONS:
Drug: Ruxolitinib cream — Ruxolitinib 1.5% cream applied twice daily.
  Other Names: INCB018424 phosphate cream

SUMMARY:
This is an open-label maximum use trial to evaluate ruxolitinib safety, tolerability and blood levels after its topical application twice daily to affected areas (≥ 35% BSA) in pediatric participants with atopic dermatitis (AD) and to determine if its systemic bioavailability results in any adverse events.

DETAILED DESCRIPTION:
Open-label, BID application to all affected areas identified at BSLN for 4 weeks (maximum use trial (MUsT) period). The next 4 weeks (treatment extension period) will be applied BID to active lesions only for the next 4 weeks for a total treatment period of 8 weeks. Eligible participants will be offered option to continue into 44-wk LTS period of BID to treat as-needed to active lesions. All participants will have 30 day safety follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children aged ≥ 2 years to < 12 years (age at the screening visit).
* Diagnosis of AD as defined by the Hanifin and Rajka (1980) criteria.
* AD duration of at least 3 months (participant/parent/guardian may verbally report signs and symptoms of AD with onset at least 3 months prior to screening).
* An IGA score as follows:

  * Treatment period: ≥ 2 at the screening and baseline visits.
  * LTS period: 0 to 4 at Week 8
* %BSA (excluding the scalp) with AD involvement as follows:

  * Treatment period: ≥ 35% at screening and baseline
  * LTS period: 0% to 20% at Week 8
* For children aged 6 years to < 12 years, mean Itch NRS score ≥ 4 during the screening period.
* Participants/guardians who agree to discontinue all agents used by the participant to treat AD from the screening visit through the final safety follow-up visit.
* At least 1 target lesion that measures approximately 5 cm2 or more at the screening and baseline visits. The target lesion must be representative of the participant's disease state but not located on the face, hands, feet, or genitalia.
* For sexually active participants, willingness to take appropriate contraceptive measures to avoid pregnancy or fathering a child for the duration of study participation with the exception of male and female participants who are prepubescent.
* Ability to comprehend and willingness to sign an ICF or written informed consent of the parent(s) or legal guardian and a verbal or written assent from the participant when possible.

Exclusion Criteria:

* An unstable course of AD (spontaneously improving or rapidly deteriorating) as determined by the investigator over the previous 4 weeks prior to the baseline visit.
* Concurrent conditions and history of other diseases as follows:

  * Immunocompromised (eg, lymphoma, acquired immunodeficiency syndrome,
  * Wiskott-Aldrich syndrome) or a history of malignant disease within 5 years before the baseline visit.
  * Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before the baseline visit.
  * Active acute bacterial, fungal, or viral skin infection (eg, herpes simplex, herpes zoster, chickenpox, clinically infected AD, impetigo) within 1 week before the baseline visit.
  * Any other concomitant skin disorder (eg, generalized erythroderma such as Netherton syndrome), pigmentation, or extensive scarring that in the opinion of the investigator may interfere with the evaluation of AD lesions or compromise participant safety.
  * Other types of eczema.
  * Chronic asthma requiring more than 800 μg/day of inhaled budesonide or equivalent high dose of other inhaled corticosteroids.
  * A medical history of hepatitis B virus or hepatitis C virus infection.
  * Any participant on maintenance dialysis.
* Any of the following clinical laboratory test results at screening:

  * Cytopenias at screening, defined as follows:
  * Hemoglobin < 10 g/dL
  * ANC < 1000/µL
  * Platelet count < 100,000/µL
  * Liver function tests:
  * AST or ALT ≥ 2.5 × ULN
  * Total bilirubin > 1.5 × ULN (isolated bilirubin > 1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin is < 35%).
  * Estimated GFR < 30 mL/min/1.73 m2 (using the Modification of Diet in Renal Disease equation)
  * Positive serology test results at screening for HIV antibody.
  * Any other clinically significant laboratory result that, in the opinion of the investigator, pose a significant risk to the participant
* Any serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, would interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* Use of any of the following treatments within the indicated washout period before the baseline visit:

  * 5 half-lives or 12 weeks, whichever is longer - biologic agents (eg, dupilumab).
  * 4 weeks - systemic corticosteroids or adrenocorticotropic hormone analogues, cyclosporine, methotrexate, azathioprine, or other systemic immunosuppressive or immunomodulating agents (eg, mycophenolate, choroquine or tacrolimus).
  * 2 weeks - immunizations with live-attenuated vaccines; sedating antihistamines unless on a long-term stable regimen (nonsedating antihistamines are permitted). Note: Live-attenuated vaccines are not recommended during the treatment period of the study. COVID-19 vaccines are allowed during the study.
  * 1 week - use of topical treatments for AD (other than bland emollients, creams, ointments, sprays, soap substitutes), topical antipruritics (eg, doxepin cream), corticosteroids, calcineurin inhibitors, PDE4 inhibitors, coal tar (shampoo), topical antibiotics, or antibacterial cleansing body wash/soap. Note: Diluted sodium hypochlorite "bleach" baths are allowed as long as they do not exceed 2 baths per week.
* Previous treatment with systemic or topical JAK inhibitors (eg, ruxolitinib, tofacitinib, baricitinib, filgotinib, lestaurtinib, pacritinib).
* Ultraviolet light therapy or prolonged exposure to natural or artificial sources of UV radiation (eg, sunlight or tanning booth) within 2 weeks prior to the baseline visit and/or intention to have such exposure during the study, which is thought by the investigator to potentially impact the participant's AD.
* Known or suspected hypersensitivity to either ruxolitinib or any component of its cream vehicle.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before the baseline visit with another investigational medication or current enrollment in another investigational drug protocol.
* Inadequate venous access in nonlesional areas for laboratory blood draws.
* In the opinion of the investigator, unable or unlikely to comply with the administration schedule and study evaluations.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events | Up to approximately 61 weeks
  Defined as any adverse event either reported for the first time or worsening of a pre-existing event after first application of study drug

SECONDARY OUTCOMES:
Concentration of Ruxolitinib in plasma | Day 1, Weeks 2, 4 and 8
Plasma Css of Ruxolitinib | Weeks 2 and 4
  Time to reach steady state concentration plateau of topical application under maximum use conditions
Accumulation ratio of Ruxilitinib | Day 1, Weeks 2, 4 and 8
  Accumulation ratio of ruxolitinib between plasma concentrations at 1 hour post application will be calculated and summarized in the age group of 7 to 11 years

CONTACTS AND LOCATIONS:
Overall Officials: Haq Nawaz, MD, MPH, MBA, MS, Study Director — Incyte Corporation
Locations (15):
- United States (15):
  - Desert Sky Dermatology, Gilbert, Arizona
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Orange County Research Center, Anaheim, California
  - Skin Care Research, Llc Scr Hollywood, Hollywood, Florida
  - Accel Clinical Research, Lake Mary, Florida
  - San Marcus Research Clinic Inc., Miami Lakes, Florida
  - Forward Clinical Trials, Tampa, Florida
  - Advanced Medical Research Pc, Sandy Springs, Georgia
  - Aeroallergy Research Lab of Savannah, Savannah, Georgia
  - Oakland Hills Dermatology Pc, Auburn Hills, Michigan
  - Skin Cancer and Dermatology Institute, Reno, Nevada
  - Forest Hills Dermatology Group, Forest Hills, New York
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Cyn3Rgy Research - Clinedge - Ppds, Gresham, Oregon
  - Progressive Clinical Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stein Gold L, Bissonnette R, Forman S, Zaenglein A, Kuo Y, Angel B, Chen X, Kallender H, Paller AS. A Maximum-Use Trial of Ruxolitinib Cream in Children Aged 2-11 Years with Moderate to Severe Atopic Dermatitis. Am J Clin Dermatol. 2025 Mar;26(2):275-289. doi: 10.1007/s40257-024-00909-5. Epub 2025 Jan 6. PMID 39760983